CLINICAL TRIAL: NCT01221909
Title: Single Dose Tranexamic Acid for Dacryocystorhinostomy
Brief Title: Tranexamic Acid in Dacryocystorhinostomy
Acronym: TA-DCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Daniel Briscoe, M.D., Chairperson of Ophthalmology Dept, EMC, Afula 18101, Israel
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: EMC-DCR-TA
Record Dates: First submitted 2010-09-18; First posted 2010-10-15 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Nasolacrimal Tract Obstruction
Keywords: bleeding; dacryocystorhinostomy; operative duration
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tranexamic acid single dose of 500mg (Experimental)
  Interventions: Drug: Tranexamic acid
- Saline (Placebo Comparator)
  Interventions: Drug: saline solution

INTERVENTIONS:
Drug: Tranexamic acid — Single dose TA 500mg or placebo will be given in DCR surgery right after the first surgical incision.
  Arms: Tranexamic acid single dose of 500mg
Drug: saline solution — 5cc saline solution
  Arms: Saline

SUMMARY:
Single dose tranexamic acid (TA) before dacryocystorhinostomy (DCR) operation: a prospective, double blind, placebo controlled study.

The study hypothesis: TA in DCR might reduce the intraoperative and postoperative bleeding in DCR surgery, and might reduce the duration of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* obstruction of nasolacrimal pathway
* eligible for DCR surgery
* 18 years of age or older

Exclusion Criteria:

* warfarin treatment
* renal insufficiency
* pregnancy
* mental retardation
* tendency to bleed
* thromboembolic disease
* thrombophilia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Duration of DCR surgery in minutes and amount of blood loss in milliliters during surgery. | Blood loss will be measured at the end of DCR operation from the suction bowel. Duration of surgery will be caculated by registering time of operation start and end.

SECONDARY OUTCOMES:
Late onset postoperative epistaxis or periorbital hematoma | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Ophthalmology, HaEmek medical center, Afula, Afula, Israel

REFERENCES:
- [Result] Ralley FE, Berta D, Binns V, Howard J, Naudie DD. One intraoperative dose of tranexamic Acid for patients having primary hip or knee arthroplasty. Clin Orthop Relat Res. 2010 Jul;468(7):1905-11. doi: 10.1007/s11999-009-1217-8. Epub 2010 Jan 9. PMID 20063079
- [Result] Wellington K, Wagstaff AJ. Tranexamic acid: a review of its use in the management of menorrhagia. Drugs. 2003;63(13):1417-33. doi: 10.2165/00003495-200363130-00008. PMID 12825966
- [Result] Astedt B. Clinical pharmacology of tranexamic acid. Scand J Gastroenterol Suppl. 1987;137:22-5. PMID 3321402